CLINICAL TRIAL: NCT03412916
Title: Integrating Mind Body Skills With Physical Activity to Improve Physical and Emotional Outcomes in Patients With Heterogeneous Chronic Pain
Brief Title: Integrating Mind-Body Skills With Physical Activity to Improve Physical and Emotional Outcomes in Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Clinical Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P000628
Record Dates: First submitted 2018-01-12; First posted 2018-01-29 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Pain; Chronic Pain; Physical Activity
Keywords: Chronic Pain; Physical Activity; Mind-body
MeSH Terms: conditions — Pain; Chronic Pain; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GetActive (Experimental): The GetActive program uses a multimodal approach to introduce and reinforce new skills, including didactics, in-session activities, discussions, and weekly practice assignments (homework). The GetActive sessions reflect a purposeful integration of the three treatment approaches (relaxation methods, stress appraisal & coping, and growth enhancement). The format is a 10-week program with weekly meetings and a focus on relaxation response strategies, cognitive behavioral training, positive psychology and mind-body interactions.
  Interventions: Behavioral: GetActive
- GetActive with Fitbit (Experimental): The GetActive with Fitbit is identical to that of the p3RP with the addition of a digital monitoring device (i.e., Fitbit) for recording of physical activity.
  Interventions: Behavioral: Get Active with Fitbit

INTERVENTIONS:
Behavioral: GetActive — GetActive is a comprehensive, multimodal treatment that was designed to increase quality of life, resiliency and ability to cope with medical symptoms and stress. This program is rooted in the elicitation of the relaxation response, a non-judgmental state of focused attention and increased awareness.
  Other Names: The Relaxation Response Resiliency Program for Pain
  Arms: GetActive
Behavioral: Get Active with Fitbit — The GetActive Program for Pain with a Digital Monitoring Device (GetActive Fitbit) is identical to the GetActive with the addition of a FitBit for recording of physical activity.
  Other Names: The Relaxation Response Resiliency Program for Pain with DMD
  Arms: GetActive with Fitbit

SUMMARY:
The aims of this study are to adapt, pilot, and examine the credibility, acceptability, and feasibility of an evidence-based mind-body program, the Relaxation Response Resiliency Program for Chronic Pain (p3RP), and the p3RP-Digital Monitoring Device (p3RP-DMD), which is the p3RP integrated with a commercial DMD, the Fitbit.

DETAILED DESCRIPTION:
The study has three phases. In phase I, the investigators are adapting the 3RP as a multidisciplinary team, and then conducting two focus groups. In phase two, the investigators are piloting the p3RP and p3RP-DMD. In phase three, the investigators are conducting a small randomized-controlled trial of the p3RP versus p3RP-DMD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age 18 years or older
* Have nonmalignant chronic pain for more than 3 months
* Able to perform a 6-minute walk test
* Owns a smartphone with Bluetooth 4.0
* Willingness and ability to participate in the 3RP intervention and to comply with the requirements of the study protocol (including weekly sessions and DMD use)
* Free of concurrent psychotropic or pain medication for at least 2 weeks prior to initiation of treatment, OR stable on current psychotropic or pain medication for a minimum of 6 weeks and willing to maintain a stable dose
* Cleared by a medical doctor for study participation
* Leads a sedentary lifestyle

Exclusion Criteria:

* Diagnosed with medical illness expected to worsen in the next 6 months
* Serious mental illness or instability for which hospitalization may be likely in the next 6 months
* Current suicidal ideation reported on self-report
* Lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder, or substance dependence
* Current substance use disorder, within the past 6 months
* Practice of yoga/meditation, or other mind-body techniques that elicit the relaxation response, once per week for 45 minutes or more within the last 3 months or less
* Regular use of DMD in the last 3 months
* Engagement in regular intensive physical exercise for >30 minute daily
* Unable to walk without use of assistance (e.g., wheelchair, walker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hopkins SW, Greenberg J, Isaacs J, Vranceanu AM. "Practice Makes Perfect"? Associations Between Home Practice and Physical and Emotional Function Outcomes Among Patients with Chronic Pain Enrolled in a Mind-Body Program. J Integr Complement Med. 2022 Apr;28(4):320-327. doi: 10.1089/jicm.2021.0324. Epub 2022 Feb 28. PMID 35231185
- [Derived] Greenberg J, Singh T, Popok PJ, Kulich RJ, Vranceanu AM. Sustainability of Improvements in Adaptive Coping Following Mind-Body and Activity Training for Chronic Pain. Int J Behav Med. 2021 Dec;28(6):820-826. doi: 10.1007/s12529-021-09971-3. Epub 2021 Mar 2. PMID 33649888
- [Derived] Greenberg J, Mace RA, Bannon SM, Kulich RJ, Vranceanu AM. Mind-Body Activity Program for Chronic Pain: Exploring Mechanisms of Improvement in Patient-Reported, Performance-Based and Ambulatory Physical Function. J Pain Res. 2021 Feb 5;14:359-368. doi: 10.2147/JPR.S298212. eCollection 2021. PMID 33574699
- [Derived] Bannon S, Greenberg J, Mace RA, Locascio JJ, Vranceanu AM. The role of social isolation in physical and emotional outcomes among patients with chronic pain. Gen Hosp Psychiatry. 2021 Mar-Apr;69:50-54. doi: 10.1016/j.genhosppsych.2021.01.009. Epub 2021 Jan 28. PMID 33540223
- [Derived] Greenberg J, Lin A, Popok PJ, Kulich RJ, Edwards RR, Vranceanu AM. Getting Active Mindfully: Rationale and Case Illustration of a Group Mind-body and Activity Program for Chronic Pain. J Clin Psychol Med Settings. 2021 Dec;28(4):706-719. doi: 10.1007/s10880-020-09758-w. Epub 2021 Jan 19. PMID 33469845
- [Derived] Greenberg J, Mace RA, Popok PJ, Kulich RJ, Patel KV, Burns JW, Somers TJ, Keefe FJ, Schatman ME, Vranceanu AM. Psychosocial Correlates of Objective, Performance-Based, and Patient-Reported Physical Function Among Patients with Heterogeneous Chronic Pain. J Pain Res. 2020 Sep 10;13:2255-2265. doi: 10.2147/JPR.S266455. eCollection 2020. PMID 32982388
- [Derived] Greenberg J, Popok PJ, Lin A, Kulich RJ, James P, Macklin EA, Millstein RA, Edwards RR, Vranceanu AM. A Mind-Body Physical Activity Program for Chronic Pain With or Without a Digital Monitoring Device: Proof-of-Concept Feasibility Randomized Controlled Trial. JMIR Form Res. 2020 Jun 8;4(6):e18703. doi: 10.2196/18703. PMID 32348281

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GetActive | GetActive With Fitbit
Started | 41 | 41
Completed | 35 | 37
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GetActive | GetActive With Fitbit | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 34 | 66
  >=65 years | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.46 (14.5) | 49.07 (14.2) | 51.77 (14.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 31 | 54
  Male | 18 | 10 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 35 | 37 | 72
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 32 | 34 | 66
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Marital status [Count of Participants; unit: Participants]
  Single, never married | 13 | 15 | 28
  Living with significant other | 5 | 6 | 11
  Married | 15 | 8 | 23
  Separated/divorced | 5 | 11 | 16
  Widowed | 3 | 1 | 4
Education [Count of Participants; unit: Participants]
  High school (12 years) | 5 | 6 | 11
  Some college/associate degree (<16 years) | 15 | 11 | 26
  Completed college (16 years) | 9 | 8 | 17
  Graduate/professional degree (>16 years) | 12 | 16 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Client Satisfaction Questionnaire 3-Item (CSQ-3) Scores Above and Below the Scale Midpoint
Description: Items are summed to generate a total score; scores range from 3 to 12, with higher values indicating higher satisfaction.
Time Frame: Post-Test (10 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 34 | 36
Participants
  Scored above the scale midpoint | 34 | 35
  Scored below the scale midpoint | 0 | 1

2. Primary Outcome: Therapist Adherence
Description: Two independent coders rated whether clinicians delivered each component of study sessions (e.g., deep breathing, providing education on prevalent myths about chronic pain) , exhibited skillful delivery (e.g., active listening, validation), and followed study protocol (e.g., collecting home practice sheets, logging attendance). Each individual component was rated on a yes/no scale. The adherent ("yes") components were summed, tallied against the total number of components in the adherence checklist, and averaged between the 2 reviewers. The score represents a total rate of adherence.
Time Frame: Collected during the intervention
Measure: Number; unit: percentage of adherence
Units Other Than Participants: Components
Arm/Group | GetActive With Fitbit | GetActive
Number analyzed (Participants) | 37 | 35
Number analyzed (Components) | 391 | 347
percentage of adherence | 94 | 98

3. Primary Outcome: Adherence to DMD - Number of Participants Who Wore DMD for ≥ 5 and < 5 Out of 7 Days
Description: Rate of participant's use of ActiGraph watch for a period of one week at both baseline and post-treatment assessments. A valid day of wear consisted of at least 7 hours of wear time.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks)
Population: The number of participants who received an ActiGraph at post-tests was fewer than baselines because of patients discontinuing participation.
Measure: Count of Participants; unit: Participants
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 33 | 39
Participants
  Baseline: Who received the ActiGraph and wore it for ≥ 5 out of 7 days | 31 | 36
  Baseline: Who received the ActiGraph and wore it for < 5 out of 7 days | 2 | 3
  Post-Test: number analyzed (Participants) | 27 | 33
  Post-Test: Who received the ActiGraph and wore it for ≥ 5 out of 7 days | 25 | 29
  Post-Test: Who received the ActiGraph and wore it for < 5 out of 7 days | 2 | 4

4. Primary Outcome: Program Safety - Number of Adverse Events Related to Study Participation
Description: Any self-reported or observed negative events related to participation.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks)
Measure: Number; unit: adverse events
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 35 | 37
adverse events | 0 | 0

5. Primary Outcome: Adherence to Home Practice - Number of Participants That Completed Homework Logs That Met Adherence Criteria
Description: Rate of participant's completion of homework assigned throughout the study. Logs were considered adherent if participants completed 3 home practice components 3 out of 7 days per week or 1 home practice component 5 out of 7 days per week.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 35 | 37
Participants
  participants that completed logs handed in met adherence criteria | 34 | 36
  participants that completed logs handed in that did not meet adherence criteria | 1 | 1

6. Primary Outcome: Feasibility of Quantitative Measures
Description: The number of participants that completed quantitative measures. Rate of participant's completion of self-report measures administered at baseline and post-test assessments.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
Participants | 41 | 40

7. Primary Outcome: Credibility and Expectancy Questionnaire (CEQ)
Description: Number of participants who score above the midpoint on two subscales assessed using frequencies and proportions. The measure involves two subscales: credibility (questions 1-3) and expectancy (questions 4-6). Subscale scores range from 3 to 27. Higher scores indicate greater perceived credibility and greater belief that treatment will help.
Time Frame: Baseline (0 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
Participants
  Expectancy: scored above the scale midpoint | 27 | 22
  Expectancy: scored below the scale midpoint | 14 | 19
  Credibility: scored above the scale midpoint | 37 | 38
  Credibility: scored below the scale midpoint | 4 | 3

8. Primary Outcome: Program Acceptability
Description: Assessed via the percentage of participants who attended at least 7 out of 10 sessions.
Time Frame: Post-Test (10 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
Participants
  Attended ≥7 out of 10 group or make-up sessions | 31 | 34
  Attended <7 out of 10 group or make-up sessions | 10 | 7

9. Secondary Outcome: 6-Min Walk Test Distance
Description: Recorded the distance in meters each participant covered by walking on a flat surface for 6 minutes.
Time Frame: 6 minutes at baseline (0 Weeks), 6 minutes at post-test (10 Weeks).
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: Meters
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
Meters
  Baseline | 346.244 (13.684) | 331.866 (13.898)
  Posttest: number analyzed (Participants) | 27 | 34
  Posttest | 389.492 (12.950) | 385.872 (12.691)

10. Secondary Outcome: ActiGraph Average Steps
Description: Average steps counted for using the wGT3X-BT ActiGraph accelerometer device. Daily step counts were collected using the device for a week at each assessment period. A weekly average was calculated from the daily totals.
Time Frame: 1 week at baseline (0 Weeks), 1 week at post-test (10 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: Steps
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 31 | 37
Steps
  Baseline | 5621.095674 (595.369) | 5226.732 (409.875)
  Posttest: number analyzed (Participants) | 26 | 30
  Posttest | 5606.226 (600.898) | 5271.760 (391.723)

11. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The PGIC assesses clinically important change in symptoms since beginning treatment. Each of the 6 items assesses a different treatment target. Items are assessed on a scale of 0 to 6. Lower scores indicate greater symptom improvement.
Time Frame: Post-Test (10 Weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 35 | 37
score on a scale
  Impression of change in pain | 2.51 (1.17) | 2.70 (1.20)
  Impression of change in physical activity | 2.31 (1.18) | 2.30 (1.10)
  Impression of change in physical function | 2.57 (1.19) | 2.78 (0.95)
  Impression of change in emotional function | 2.40 (1.01) | 2.54 (0.84)
  Impression of change in resiliency | 2.14 (0.91) | 2.32 (1.03)
  Impression of change from use of Fitbit | NA (NA) | 1.86 (0.95)

12. Secondary Outcome: Physical Activity Scale for Persons With Physical Disabilities (PASIPD)
Description: The PASIPD is a 13-item measure that assesses one's level of physical activity and exercise in the past 7 days. Scores range from 0 to 100. Higher scores indicate greater activity.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), 3-Month Follow-Up (23 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
score on a scale
  Baseline | 9.200 (1.073) | 14.213 (2.819)
  Posttest: number analyzed (Participants) | 35 | 37
  Posttest | 10.985 (1.422) | 16.742 (2.421)
  Follow up: number analyzed (Participants) | 28 | 29
  Follow up | 9.097 (1.280) | 13.396 (1.791)

13. Secondary Outcome: WHO Disability Assessment Schedule 2.0 (WHODAS)
Description: The WHODAS measures level of functioning in six domains: cognition, mobility, self-care, getting along, life activities, and participation. Scores range from 0 to 100. Higher scores indicate more disability.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), 3-Month Follow-Up (23 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
score on a scale
  Baseline | 26.91 (2.51) | 36.64 (3.28)
  Posttest: number analyzed (Participants) | 35 | 37
  Posttest | 18.56 (2.28) | 27.88 (2.71)
  Follow-up: number analyzed (Participants) | 28 | 29
  Follow-up | 20.88 (3.17) | 27.42 (3.38)

14. Secondary Outcome: Patient-Reported Outcomes Measurement Information System Physical Function v.8b
Description: The 8-item scale assesses for how difficult it is for one to perform daily living activities. Raw scores range from 8 to 40. T scores range from 20.3 to 60.1. Higher scores indicate better physical function and ability to perform activities of daily living.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), 3-Month Follow-Up (23 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
score on a scale
  Baseline | 39.74 (1.05) | 37.29 (1.26)
  Posttest: number analyzed (Participants) | 35 | 37
  Posttest | 42.27 (1.21) | 40.18 (1.37)
  Follow-up: number analyzed (Participants) | 28 | 29
  Follow-up | 44.70 (1.35) | 41.30 (1.65)

15. Secondary Outcome: Patient-Reported Outcomes Measurement Information System Anxiety v.8a
Description: The 8-item scale measures fear and worry over the past week. Raw scores range from 8 to 40. T-scores range from 37.1 to 83.1. Higher scores indicate higher levels of anxiety.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), 3-Month Follow-Up (23 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
score on a scale
  Baseline | 53.50 (1.58) | 59.33 (1.39)
  Posttest: number analyzed (Participants) | 35 | 37
  Posttest | 51.26 (1.41) | 56.39 (1.53)
  Follow-up: number analyzed (Participants) | 28 | 29
  Follow-up | 51.49 (1.68) | 57.27 (1.62)

16. Secondary Outcome: Patient-Reported Outcomes Measurement Information System Depression v.8b
Description: The 8-item scale measures depressive symptoms over the past week. Raw scores range from 8 to 40 and t scores range from 37.1 to 82.4. Higher scores indicate greater depressive symptoms.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), 3-Month Follow-Up (23 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
score on a scale
  Baseline | 53.14 (1.69) | 60.02 (1.45)
  Posttest: number analyzed (Participants) | 35 | 37
  Posttest | 50.21 (1.55) | 55.74 (1.21)
  Follow-up: number analyzed (Participants) | 28 | 29
  Follow-up | 50.21 (1.54) | 55.75 (1.70)

17. Secondary Outcome: Pain Resilience Scale (PRS)
Description: The PRS, a 14-item scale, measures pain resilience and how one would respond emotionally when faced with prolonged pain. Scores range from 0 to 56. Higher scores indicate greater resilience.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), 3-Month Follow-Up (23 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
score on a scale
  Baseline Pain resilience | 37.68 (1.47) | 32.51 (1.58)
  Posttest Pain resilience: number analyzed (Participants) | 35 | 37
  Posttest Pain resilience | 43.55 (1.64) | 36.19 (1.82)
  3-Month follow- up Pain resilience: number analyzed (Participants) | 28 | 29
  3-Month follow- up Pain resilience | 45.02 (1.39) | 36.13 (2.07)

18. Secondary Outcome: Numerical Rating Scale
Description: Measures pain at rest and pain with activity on a Likert scale with 0 being no pain and 10 being the worst pain ever
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), 3-Month Follow-Up (23 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
score on a scale
  Baseline Pain at rest | 5.07 (0.39) | 5.70 (0.34)
  Posttest Pain at rest: number analyzed (Participants) | 35 | 37
  Posttest Pain at rest | 3.73 (0.41) | 4.58 (0.36)
  Follow up Pain at rest: number analyzed (Participants) | 28 | 29
  Follow up Pain at rest | 4.18 (0.41) | 4.30 (0.50)
  Baseline Pain during activity | 6.93 (0.31) | 7.15 (0.34)
  Posttest Pain during activity: number analyzed (Participants) | 35 | 37
  Posttest Pain during activity | 5.16 (0.42) | 6.01 (0.41)
  Follow-up Pain during activity: number analyzed (Participants) | 28 | 29
  Follow-up Pain during activity | 5.28 (0.45) | 5.31 (0.60)

19. Secondary Outcome: Cognitive and Affective Mindfulness Scale (CAMS)
Description: The CAMS, a 12-item scale, measures how much one experiences their thoughts and feelings. Items range from 1 to 4. Total scores range from 12 to 48. Higher values reflect higher levels of mindfulness.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), 3-Month Follow-Up (23 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
score on a scale
  Baseline Mindfulness | 32.12 (0.99) | 30.29 (1.11)
  Posttest Mindfulness: number analyzed (Participants) | 35 | 37
  Posttest Mindfulness | 36.09 (1.07) | 33.07 (1.00)
  Three-Month follow-up Mindfulness: number analyzed (Participants) | 28 | 29
  Three-Month follow-up Mindfulness | 35.95 (1.09) | 34.08 (1.36)

20. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: Measures one's sleep quality. Scores range from 0 to 21. Higher scores indicate worse sleep quality.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), 3-Month Follow-Up (23 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
score on a scale
  Baseline | 8.756 (.664) | 11.293 (.629)
  Post-test: number analyzed (Participants) | 35 | 37
  Post-test | 6.979 (.622) | 10.754 (.686)
  Follow up: number analyzed (Participants) | 28 | 29
  Follow up | 6.565 (.558) | 10.046 (.737)

21. Secondary Outcome: Patient-Reported Outcomes Measurement Information System Social Isolation v.4a
Description: The 4-item scale measures how often one perceives feeling apart from others and excluded. Raw scores range from 4 to 20. Scaled scores range from 34.8 to 74.2. Higher scores indicate greater social isolation.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), 3-Month Follow-Up (23 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- GetActive-Fitbit: The GetActive with Fitbit is identical to that of the p3RP with the addition of a digital monitoring device (i.e., Fitbit) for recording of physical activity.
  Get Active with Fitbit: The GetActive Program for Pain with a Digital Monitoring Device (GetActive Fitbit) is identical to the GetActive with the addition of a FitBit for recording of physical activity.
Arm/Group | GetActive | GetActive-Fitbit
Number analyzed (Participants) | 41 | 41
score on a scale
  Baseline | 48.788 (1.743) | 51.880 (1.538)
  Post-test: number analyzed (Participants) | 35 | 37
  Post-test | 45.364 (1.556) | 49.793 (1.629)
  Follow-up: number analyzed (Participants) | 28 | 29
  Follow-up | 47.582 (1.673) | 51.252 (1.916)

22. Secondary Outcome: Patient-Reported Outcomes Measurement Information System Emotional Support v.4a
Description: The 4-item scale measures perceived emotional support. Raw scores range from 4 to 20. Scaled scores range from 25.7 to 62. Higher score indicate greater emotional support.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), 3-Month Follow-Up (23 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
score on a scale
  Baseline | 49.924 (1.365) | 48.432 (1.288)
  Post-test: number analyzed (Participants) | 35 | 37
  Post-test | 53.078 (1.604) | 50.330 (1.560)
  Follow-up: number analyzed (Participants) | 28 | 29
  Follow-up | 53.425 (1.417) | 52.311 (1.845)

23. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: The PCS, a 13-item scale, measures how individuals experience pain, in terms of catastrophizing. Total scores range from 0 to 52. A higher score indicates more catastrophizing.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), 3-Month Follow-Up (23 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
score on a scale
  Baseline | 19.71 (1.84) | 22.27 (1.89)
  Posttest: number analyzed (Participants) | 35 | 37
  Posttest | 9.98 (1.29) | 16.75 (1.77)
  Three-Month follow-up: number analyzed (Participants) | 28 | 29
  Three-Month follow-up | 9.91 (1.49) | 16.79 (2.03)

24. Secondary Outcome: Tampa Kinesiophobia Scale (TKS)
Description: The TKS is a 17-item scale that measures one's fear of movement, with a greater score indicating greater fear of injury due to movement. Scores range from 11 to 44.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), 3-Month Follow-Up (23 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
score on a scale
  Baseline | 38.65 (1.32) | 39.54 (1.38)
  Posttest: number analyzed (Participants) | 35 | 37
  Posttest | 31.42 (1.27) | 35.22 (1.32)
  3-Month follow- up: number analyzed (Participants) | 28 | 29
  3-Month follow- up | 35.82 (1.46) | 35.92 (1.45)

25. Secondary Outcome: Measure of Current Status (MOCS-A)
Description: The MOCS-A, a 13-item scale, measures one's perceived ability to perform various skills that the intervention aims to target. Scores range from 0 to 52. Higher scores indicate greater perceived ability.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), 3-Month Follow-Up (23 Weeks)
Population: We used linear mixed-models repeated measures analyses of covariance, which implicitly impute unobserved data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | GetActive | GetActive With Fitbit
Number analyzed (Participants) | 41 | 41
score on a scale
  Baseline Adaptive Coping | 27.56 (1.49) | 27.27 (1.50)
  Posttest Adaptive Coping: number analyzed (Participants) | 35 | 37
  Posttest Adaptive Coping | 36.09 (1.43) | 34.10 (1.33)
  Three-Month follow-up Adaptive Coping: number analyzed (Participants) | 28 | 29
  Three-Month follow-up Adaptive Coping | 34.24 (1.50) | 31.98 (1.36)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | GetActive | GetActive With Fitbit
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/37
Serious Adverse Events (participants affected / at risk) | 1/35 | 1/37
Other Adverse Events (participants affected / at risk) | 3/35 | 7/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GetActive (N=35) | GetActive With Fitbit (N=37)
Stroke (Vascular disorders) | 1 | 0
Fall (Musculoskeletal and connective tissue disorders) | 0 | 1 — Patient admitted to hospital; suffered falls; celluitis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GetActive (N=35) | GetActive With Fitbit (N=37)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Sprained quadricep muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain Flare (Musculoskeletal and connective tissue disorders) | 1 | 1
Sickle Cell Anemia Flare (Blood and lymphatic system disorders) | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 0 | 1 — Patient hospitalized for diverticulitis attack
Chemotherapy (Surgical and medical procedures) | 0 | 1 — Patient hospitalized for chemotherapy
Hospitalization (General disorders) | 0 | 1 — Patient admitted to the hospital for unknown reasons.
Elevated blood pressure and heart rate (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT03412916/Prot_SAP_000.pdf